CLINICAL TRIAL: NCT05149833
Title: An Observational Study of Diagnostic Criteria, Clinical Features and Management of Opioid Induced Constipation (OIC) in European Patients With Cancer Pain
Brief Title: European Study of Opioid Induced Constipation
Acronym: E-StOIC
Status: Completed | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Prof Andrew Davies, Professor of Palliative Medicine, University of Dublin, Trinity College
Other Study IDs: PM2021/65
Record Dates: First submitted 2021-10-05; First posted 2021-12-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Opioid-Induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Constipation is common (40-90%) in advanced cancer patients , and has a significant negative impact on quality of life. The aetiology of constipation is often multifactorial in advanced cancer patients. However, it is well recognised that opioid analgesics are a common cause of constipation in this group. The prevalence of opioid-induced constipation (OIC) is stated to be 40-70%, although a recent large study reported an even higher figure.

OIC has been reported to exceed pain in terms of distress caused, and studies have found that some patients choose to reduce or discontinue opioid medication in order to attempt to better control constipation. Moreover, OIC is associated with a variety of physical (gastrointestinal, systemic), psychological and social problems.

DETAILED DESCRIPTION:
This European study follows on from a United Kingdom study, and aims to confirm findings of the previous study in a larger, more heterogeneous sample: it also aims to explore additional strategies to manage OIC. Moreover, the study aims to identify differences in perception of normal bowel habit / constipation, and differences in OIC management in the different European countries. Previous studies suggest that there are cultural differences in people's beliefs about constipation / normal bowel function. The aim of the project is to investigate OIC in a real world / heterogenous group of European patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Diagnosis of cancer
* Diagnosis of cancer pain or cancer treatment-related pain
* Taking regular opioids for at least one week (i.e. opioid for mild to moderate pain / "weak" opioid; or opioid for moderate to severe pain / "strong" opioid)

Exclusion Criteria:

* Unable to provide consent
* Unable to complete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants may be inpatients, or outpatients at the study sites. Participants must meet all of the inclusion criteria for the study, and none of the exclusion criteria for the study. Participants must have a diagnosis of cancer and be on regular opioids for at least one week for cancer/ cancer treatment related pain.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of opioid induced constipation (OIC) | 5 minutes
  OIC diagnosed using Rome IV diagnostic criteria

SECONDARY OUTCOMES:
Impact of OIC on quality of life | 5 minutes
  Patient Assessment of Constipation Quality of Life tool score Scale 0-4 (better to worse)
Efficacy of treatment for OIC | 3 minutes
  Bowel Function Index tool score Score 0-100 (better to worse)
Adherence with treatment for OIC No scale - yes / no options | 5 minutes
  Study questionnaire
Use of non-prescribed treatments for OIC | 5 minutes
  Study questionnaire No scale - yes / no options

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, MD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Norah Fagan, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fallon MT, Hanks GW. Morphine, constipation and performance status in advanced cancer patients. Palliat Med. 1999 Mar;13(2):159-60. doi: 10.1191/026921699677653615. No abstract available. PMID 10474699
- [Background] Goodman M, Low J, Wilkinson S. Constipation management in palliative care: a survey of practices in the United kingdom. J Pain Symptom Manage. 2005 Mar;29(3):238-44. doi: 10.1016/j.jpainsymman.2004.06.013. PMID 15781174
- [Background] van den Beuken-van Everdingen MH, de Rijke JM, Kessels AG, Schouten HC, van Kleef M, Patijn J. Quality of life and non-pain symptoms in patients with cancer. J Pain Symptom Manage. 2009 Aug;38(2):216-33. doi: 10.1016/j.jpainsymman.2008.08.014. Epub 2009 Jun 28. PMID 19564094
- [Background] Cherny N, Ripamonti C, Pereira J, Davis C, Fallon M, McQuay H, Mercadante S, Pasternak G, Ventafridda V; Expert Working Group of the European Association of Palliative Care Network. Strategies to manage the adverse effects of oral morphine: an evidence-based report. J Clin Oncol. 2001 May 1;19(9):2542-54. doi: 10.1200/JCO.2001.19.9.2542. PMID 11331334
- [Background] Davies A, Leach C, Butler C, Gregory A, Henshaw S, Minton O, Shorthose K, Batsari KM. Opioid-induced constipation in patients with cancer: a "real-world," multicentre, observational study of diagnostic criteria and clinical features. Pain. 2021 Jan;162(1):309-318. doi: 10.1097/j.pain.0000000000002024. PMID 32701649
- [Background] Walter S, Hallbook O, Gotthard R, Bergmark M, Sjodahl R. A population-based study on bowel habits in a Swedish community: prevalence of faecal incontinence and constipation. Scand J Gastroenterol. 2002 Aug;37(8):911-6. doi: 10.1080/003655202760230865. PMID 12229965
- [Background] Lee TH, Choi SC, Park MI, Park KS, Shin JE, Kim SE, Jung KW, Koo HS, Kim WJ, Cho YK, Kim YS, Lee JS. Constipation misperception is associated with gender, marital status, treatment utilization and constipation symptoms experienced. J Neurogastroenterol Motil. 2014 Jul 31;20(3):379-87. doi: 10.5056/jnm14011. PMID 24935009
- [Derived] Davies A, Fagan N, Power J, Taylor A. 'Constipation': One word, many meanings amongst persons with cancer: An observational study. Palliat Med. 2025 May;39(5):553-562. doi: 10.1177/02692163251325711. Epub 2025 Mar 12. PMID 40071858